CLINICAL TRIAL: NCT07120919
Title: The Effect of Peer Education on Reproductive Health and Safe Sexuality Knowledge Level: A Randomised Controlled Experimental Study
Brief Title: Effect of Peer Education on Reproductive Health and Safe Sexuality Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, EMİNE AVCU, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025/177
Record Dates: First submitted 2025-07-23; First posted 2025-08-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-04

CONDITIONS: Knowledge Level
Keywords: peer education; reproductive health education; family planning education; impact of peer education

STUDY DESIGN:
Intervention Model Description: randomised controlled experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEER EDUCATION (Experimental): Safe sexuality and reproductive health trainings for young people by peer mentors.
  Interventions: Other: Peer Educatıon
- BROCHURE (No Intervention): Providing only a training brochure without any intervention

INTERVENTIONS:
Other: Peer Educatıon — The peer educators provided training on reproductive health and safe sexuality for young people and completed the intervention part by giving training brochures to the participants.
  Arms: PEER EDUCATION

SUMMARY:
The aim of this study is to examine the effect of Safe Sexuality and Family Planning Education with Peer Education on Midwifery Students, to create awareness on this issue and to contribute to the literature. The main questions aimed to be answered in the study are as follows:

H1: The level of reproductive health knowledge of students receiving peer education is significantly higher than the control group who did not receive education.

H2: The safe sexuality knowledge level of students receiving peer education is significantly higher than the control group who did not receive education.

H3: Peer education provides a statistically significant increase in students' overall reproductive health and safe sex knowledge levels.

Participants will evaluate the training with the scales they will fill in before and after the safe sexuality and family planning training. also, the effect of the training on behaviour will be measured with the questionnaires they will fill in 2 months later.

DETAILED DESCRIPTION:
The study population consisted of Turkish midwifery students studying at Istanbul Medipol University, Faculty of Health Sciences, in the 1st, 2nd, 3rd, and 4th grades. The sample of the study was determined by stratified random sampling among Turkish students. Students who agreed to participate in the study were assigned to intervention and control groups by the lottery method. The number of students participating in the study by class was as follows:

1. st year: 25 intervention, 25 control,
2. nd year: 31 intervention, 31 control,
3. rd year: 18 intervention, 18 control,
4. th year: 26 intervention, 26 control.

Inclusion Criteria:

At least 18 years old,

Being a midwifery student,

Able to communicate verbally,

Volunteering to participate in the study.

Exclusion Criteria:

History of psychiatric illness,

Being a foreign national student.

Data Collection Tools: The study data were collected using the Participant Information Form, "Reproductive Health Scale for Turkish Adolescents," and "Peer Mentoring Evaluation Scale."

Participant Information Form: This form consisted of 15 questions developed by the researchers in line with the literature.

Reproductive Health Scale for Turkish Adolescents: This 34-item scale was in a 5-point Likert type format. The first 16 items were reverse-scored. The Cronbach's alpha coefficient of the scale was 0.88.

Peer Mentoring Evaluation Scale: Developed by Kocadere in 2015, the scale consisted of 10 items in a 7-point Likert type format. A total peer mentoring score was obtained by summing all responses. The minimum possible score was 10, and the maximum was 70. Higher total scores indicated higher satisfaction. The Cronbach's alpha coefficient of the scale was 0.937.

Data Collection:

Data were collected via Google survey. The Google survey link of the data collection tools was shared with the students, and the informed consent form was obtained face-to-face. The online questionnaire form was set to be answered only from a single account to prevent multiple responses from the same participant. Students who volunteered to participate read the study information and clicked the confirmation tab to join the study. It took approximately 15 minutes for participants to complete the survey.

The peer educators were selected as two volunteer participants from the "Reproductive Health Peer Clinic" project of the Midwifery Department at Istanbul Medipol University, and their names were recorded in the study's ethics committee form. The "Reproductive Health Peer Clinic" project was supported by the Social Contribution Commission of Istanbul Medipol University. Within the scope of the project, a room in the Midwifery Department was transformed into a clinic, and final-year midwifery students provided counseling on reproductive health and family planning to all university students. The Turkish Family Planning Association was a stakeholder in this project and organized the orientation of peer educators. Counseling was provided by midwifery students three days a week, and gynecological examinations were offered free of charge one day a week. Peer educators were chosen from final-year midwifery students because they had completed all core theoretical courses, had strong scientific knowledge, and were gaining professional experience through clinical practice three days a week. The privacy of student clients was protected, and their data were kept confidential. In the training conducted within the study, brochures on contraceptive methods and safe sexuality for young people, prepared by peer educators, were used.

In the intervention group, the "Reproductive Health Scale for Turkish Adolescents" was administered in the pre-test, and safe sexuality and youth-focused safe sexuality training was provided along with brochures. Three months later, in the post-test, both the "Reproductive Health Scale for Turkish Adolescents" and the "Peer Mentoring Evaluation Scale" were administered. In the control group, no intervention was performed, and only brochures were given along with the administration of the "Reproductive Health Scale for Turkish Adolescents."

Data Analysis:

The data obtained in the study were analyzed using SPSS version 25.0. First, the normality of the variables was assessed, and appropriate statistical tests were selected accordingly. For comparisons between groups of quantitative data, the Independent Samples t-test was used; for data not conforming to normal distribution, Mann-Whitney U or Wilcoxon tests were preferred. Cohen's d effect size analysis was performed to determine the magnitude of significant differences. Additionally, the Independent Samples t-test was used to compare the means of two independent groups, the Paired Samples t-test to compare the means of the same group at two different time points, the Chi-square test to examine the relationship between two categorical variables, One-Way ANOVA to compare the means of three or more groups, and Two-Way ANOVA to examine the effect of two independent variables and their interaction. The level of significance was set at p<0.05 in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old,
* Midwifery student,
* Can communicate verbally,
* Volunteer to participate in the research.

Exclusion Criteria:

* Has a history of psychiatric illness.
* Foreign students.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It was applied to midwifery students and since men are not accepted to the midwifery department in Turkey, it was applied to women.
Enrollment: 200 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Reproductive Health Scale for Turkish Adolescents | baseline
  The scale, which was developed to measure the level of knowledge of young people about reproductive health and consists of 34 items, is 5-point Likert type. The first 16 items are reverse scored. Cronbach's alpha=0.88.

SECONDARY OUTCOMES:
Peer Mentoring Assessment Scale | 3 months later.
  The scale consists of 10 items. In the 7 Likert scale, a total score for peer mentoring is obtained by summing all responses. The lowest total score is 10 and the highest score is 70. The higher the total score, the higher the satisfaction. The scale has α = 0.937.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, BEYKOZ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected during this study will not be shared with other researchers due to privacy concerns and institutional policies.